CLINICAL TRIAL: NCT00300820
Title: Seeking Genetic Counseling: What Motivates Families At Risk For Psychiatric Illness?
Brief Title: Perspectives of Individuals With Bipolar Disorder and Siblings of Individuals With Bipolar Disorder; A Telephone Interview Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060108; 06-HG-0108
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-02-06

CONDITIONS: Bipolar Disorder (BD); Bipolar
Keywords: Bipolar Disorder; Affected Adults and Adult Siblings; Interest in Genetic Counseling; Bipolar; Genes; Familial; Education; Testing; BP; Adult Siblings
MeSH Terms: conditions — Bipolar Disorder

SUMMARY:
This study will examine those who will seek and those who are most likely to benefit from genetic counseling for psychiatric disorders. It will identify themes related to perceived risks, benefits, and possible motivations for seeking genetic counseling among families affected by bipolar disorder. It will then use those themes to generate a starting point for a framework to guide further research and to improve genetics services as they are currently practiced.

Adults with bipolar disorder and the adult siblings of people with bipolar disorder are eligible for this study. In a 60- to 90-minute telephone interview, participants are asked questions related to their thoughts about the causes of bipolar disorder, their experiences with the illness, their concerns about the disorder occurring again in their families, and their feelings about the value of discussing these issues with health care professionals. They also are asked questions about the mental health of their close family members and their own mental health.

DETAILED DESCRIPTION:
This study aims to examine through the use of qualitative telephone interviews who will seek, and who is most likely to benefit from, genetic counseling for psychiatric disorders. The specific aims are to identify themes related to perceived risks, benefits, and possible motivations for seeking genetic counseling among families affected by bipolar disorder; to use those themes to generate a starting point for a conceptual framework to guide further research; and to use those themes to improve clinical genetics services currently in practice.

None of the few available studies on genetics and bipolar disorder evaluate interest in genetic services in the absence of genetic testing (e.g., family-history-based risk assessment, education about etiology, psychological support) even though those elements will continue to be relevant even if genetic testing becomes available. Only one study asked any questions about psychiatric genetic counseling in the absence of testing-a study on schizophrenia in which one such question was posed. In most of the available literature, the focus is on highly predictive testing scenarios that are not relevant in current practice, and may never be relevant. In addition, most studies test the researchers' preconceived notions of risks and benefits, without allowing participant input. More research will facilitate the integration of genetic counseling for psychiatric disorders into the genetics clinic.

This is a qualitative study using telephone interviews that will be taped and transcribed. We plan to interview 15 to 25 adults affected with bipolar disorder and 15 to 25 unaffected adult siblings. We will use a semi-structured interview guide that will allow the integration of new elements and the modification of existing elements. We will use data reduction and coding to synthesize the most important themes.

This study will result in themes that can be tested in a larger, more representative sample, allowing us to test hypotheses about interest in psychiatric genetic counseling. This study also will provide preliminary data about anticipating, through the use of realistic scenarios, the point at which individuals are more likely to embrace psychiatric genetic counseling; and beginning to understand, in a broader perspective, what may increase or decrease interest in genetic counseling and risk assessment based on family history for complex disorders. More immediately, this study will provide a description of the experience of living with risk in the family that should be of interest to genetics professionals.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals over 18 years of age who have been diagnosed with bipolar disorder (per their own report; no screening will be performed), and/or the adult siblings of affected individuals. Participants do not have to be sibling pairs, i.e., an affected individual may be included without the participation of their unaffected sibling, and visa versa. Participants must be able to speak English fluently.

EXCLUSION CRITERIA:

Those under 18 years of age will not be included. First-degree relatives other than full siblings will not be included. If a participant is symptomatic to the point that the interview is compromised, as determined by the PI who has considerable experience counseling affected individuals, the PI will end the interview and any data collected will be destroyed. If possible, the interview will be rescheduled. We will encourage symptomatic individuals to seek care from their mental health provider, or we will make a referral if the individual does not have a provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-03-02; Study Completion 2008-02-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hodgkinson KA, Murphy J, O'Neill S, Brzustowicz L, Bassett AS. Genetic counselling for schizophrenia in the era of molecular genetics. Can J Psychiatry. 2001 Mar;46(2):123-30. doi: 10.1177/070674370104600202. PMID 11280080